CLINICAL TRIAL: NCT06358560
Title: Applied Clinical Neuroscience and Its Effect on Self-reported Stress and Other Physiological Markers
Status: Recruiting | Type: Observational
Sponsor: Dylan Saulsbery (Other)
Responsible Party: Sponsor-Investigator, Dylan Saulsbery, Director, The Brain Health Clinics
Organization: The Brain Health Clinics (Other)
Other Study IDs: BrainHealthClinics
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Stress
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Therapeutic exercises — Rehabilitation exercises designed to achieve the treatment goal

SUMMARY:
The purpose of this study is to see if an applied clinical neuroscience (ACN) approach to the symptom of 'stress' has a measurable effect on an individual's self-reported stress level. Physiological markers will be measured and analyzed to potentially allow for greater insight and aid in setting up any future research on this topic. This is an independent research study.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must be presenting to the clinic for treatment for 'stress'.

Exclusion Criteria:

* Under 18 years of age
* No vulnerable populations (physical or mental disability, economically or educationally disadvantaged, pregnancy, minors, persons incarcerated).
* No participants that have an additional relationship beyond the doctor/patient relationship that exists by nature of a patient committing to treatment (a family member or clinic employee would be excluded from the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit the first 5-15 people that present to the clinic on their own for treatment for 'stress'.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox® Item Bank v3.0 - Perceived Stress (Ages 18+) - Fixed Form | through study completion, an average of 6 months
  There are 10 questions that are answered on a scale of 1-5, for a final score ranging from 10-50. The higher the number the worse the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Brain Health Clinics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided